CLINICAL TRIAL: NCT06955039
Title: Effects of Sand Exercise Program On Foot Posture , Navicular Drop and Dynamic Balance in Children With Pronated Foot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC//RER/AHS/24/0733
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Pronated Foot
Keywords: Pronated foot; sand exercise program; navicular drop; foot posture

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial (RCT) perfomed in which 20 participants divided into 2 groups an experimental group and a control group to assess the effects of an 8-week exercise program on foot health in children with pronated feet. The experimental group will perform sand activities and towel curl exercises three times a week, while the control group will only perform towel curl exercises. Pre values were taken at 1st week and then after 4th week mid values of interventions will be taken and post values of intervention will be taken after 8th week of intervention to measure foot posture, navicular drop, and dynamic balance using the Foot Posture Index (FPI-6), Navicular Drop Test, Y Balance Test, and Feiss Line Test.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Clinical experimental: For group A each session last 50 minutes daily for 8 weeks 3 times per week during a 8-week period
  Interventions: Other: Sand Activites; Other: Towel Curl Exercises; Other: (TCE)
- Group B (Active Comparator): Clinical experimental: For group B each session lasted for 5 minutes. The exercise was performed in three sets per week, with each set lasting 5 minutes. Participants performed the exercise 20-25 times for 8 weeks
  Interventions: Other: Sand Activites; Other: Towel Curl Exercises; Other: (TCE)

INTERVENTIONS:
Other: Sand Activites — Exercises included walking, jogging, striding, bounding, galloping, and short sprints.Exercise intensity (running speed) was controlled using a stopwatch and predefined running distances on the sand-based exercise court.
Other: Towel Curl Exercises — The experimental group will perform Towel Curl Exercises Sand .In Week 1-4 the exercises will conducted without weights while in weeks 5-8 the exercise included the use of dumbbells weighing 2kg.this exercises will conducted in a sitting position on a slick surface.
Other: (TCE) — The control group will only perform towel curl exercises In Week 1-4 the exercises will conducted without weights while in weeks 5-8 the exercise included the use of dumbbells weighing 2kg.this exercises will conducted in a sitting position on a slick surface.

SUMMARY:
This randomized controlled trial investigates the effects of combining sand training with navicular drop interventions on foot posture and dynamic balance in children aged 6-11 with pronated feet. Pronated foot posture, marked by inward foot rolling and a lowered arch, can impair gait and balance. Early intervention is key to preventing long-term issues. Twenty participants will be divided into experimental and control groups. Over eight weeks, the experimental group will perform sand and towel curl exercises, while the control group will do towel curls only. Foot posture, navicular drop, and balance will be assessed using the FPI-6, Navicular Drop Test, Y Balance Test, and Feiss Line Test at baseline, 4 weeks, and 8 weeks. The study aims to evaluate the added benefits of sand training in improving pediatric foot health.

DETAILED DESCRIPTION:
The effects of sand training exercises combined with navicular drop interventions on dynamic balance and foot posture in children aged 6 to 11 years with pronated feet. Pronated foot posture, characterized by the inward rolling of the foot and a lowered medial arch, is prevalent in pediatric populations and can lead to altered gait mechanics and reduced dynamic balance. Early intervention is crucial to prevent long-term deformities and improve overall foot health. The study aims to provide evidence-based insights into the benefits of integrating proprioceptive training with specific sand exercises program targeting the navicular bone, thereby enhancing foot posture and dynamic balance in affected children.

This randomized controlled trial (RCT) will involve 20 participants divided into an experimental group and a control group to assess the effects of an 8-week exercise program on foot health in children with pronated feet. The experimental group will perform sand activities and towel curl exercises three times a week, while the control group will only perform towel curl exercises. The study will measure foot posture, navicular drop, and dynamic balance using the Foot Posture Index (FPI-6), Navicular Drop Test, Y Balance Test, and Feiss Line Test, with assessments conducted at baseline, 4 weeks, and 8 weeks post-intervention. This study aims to provide evidence on the effects of combining sand training with towel curl exercises for determining foot posture.

ELIGIBILITY:
Inclusion Criteria:

* Children aged [6-11] years with bilateral pronated feet.
* Both gender
* No recent foot injury or lower extremity pain from last six months
* Has no history of foot and ankle surgery lifetime
* All eligible children were assessed with the Feiss line method

Exclusion Criteria:

* the presence of pain in the foot at the time of physical examination
* injury to the lower limbs, such as musculoskeletal injuries, during the previous 6 months congenital structural abnormalities, cerebral palsy, motor dysfunction prior surgery affecting the foot

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-06-17 (Estimated); Study Completion 2025-06-18 (Estimated)

PRIMARY OUTCOMES:
Feiss line Test | base line ,4th week ,8th week
  The Feiss Line Test assesses the medial longitudinal arch by drawing a line from the medial malleolus to the first metatarsophalangeal joint. The navicular tuberosity should lie on or near this line; displacement below indicates arch lowering. A perpendicular distance from the navicular to this line is measured-positive if above, negative if below. The test shows high reliability, with inter-tester ICC of 0.94 and intra-tester ICC of 0.91, indicating consistent measurements across and within testers.
Foot Posture Index (FPI -6 ) | base line ,4th week ,8th week
  Foot posture is assessed using the Foot Posture Index (FPI-6) with the subject barefoot in a relaxed standing position. It evaluates six criteria across the forefoot, midfoot, and hindfoot, including talar head palpation, malleolar curvature, calcaneal position, talonavicular prominence, medial arch height, and forefoot alignment. Scores range from -12 (highly supinated) to +12 (highly pronated). The FPI-6 is a quick, simple, and reliable tool, showing strong intra-rater reliability (ICC 0.81-0.92) and good inter-rater reliability (ICC 0.69), especially in pediatric assessments.
Navicular Drop Measurement | base line ,4th week ,8th week
  The Navicular Drop Test (NDT) measures foot pronation by comparing navicular height in a seated subtalar neutral position to its height in relaxed standing. It shows moderate to good intra-rater reliability, with ICC values ranging from 0.61 to 0.79, making it a useful clinical tool for assessing pronation
Dynamic Balance Assessment | base line ,4th week ,8th week
  The Star Balance Test (or Y-Balance Test) assesses dynamic balance by having participants reach in three directions-anterior, posteromedial, and posterolateral-while balancing on one foot. The test is performed clockwise for the right foot and counterclockwise for the left. Reach distance is recorded, and errors require a retest. It shows good interrater reliability with ICC values of 0.80-0.85 and a standard error of 3.1-4.2 cm.

CONTACTS AND LOCATIONS:
Overall Officials: Eishah M Saeed, MS-PPT, Principal Investigator — Riphah International University
Locations (1):
- Rising Sun Institute, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alam F, Raza S, Moiz JA, Bhati P, Anwer S, Alghadir A. Effects of selective strengthening of tibialis posterior and stretching of iliopsoas on navicular drop, dynamic balance, and lower limb muscle activity in pronated feet: A randomized clinical trial. Phys Sportsmed. 2019 Sep;47(3):301-311. doi: 10.1080/00913847.2018.1553466. Epub 2018 Dec 5. PMID 30517043